CLINICAL TRIAL: NCT01347385
Title: Barbed Suture Versus Traditional Suture Material for Laparoscopic Myomectomy: A Randomized Controlled Trial
Brief Title: Barbed Suture Versus Traditional Suture Material for Laparoscopic Myomectomy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sunnybrook Health Sciences Centre (Other)
Responsible Party: Jamie Kroft, MD, FRCSC, Sunnybrook Health Sciences Centre, University of Toronto
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MIS-1
Record Dates: First submitted 2011-04-26; First posted 2011-05-04 (Estimated); Last update posted 2011-05-04 (Estimated); Status verified 2011-04

CONDITIONS: Fibroids
Keywords: Fibroids; Laparoscopic myomectomy; Barbed suture
MeSH Terms: conditions — Leiomyoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Barbed suture (Experimental)
  Interventions: Procedure: Laparoscopic myomectomy with unidirectional barbed suture
- Traditional suture material (Active Comparator)
  Interventions: Procedure: Traditional suture material

INTERVENTIONS:
Procedure: Laparoscopic myomectomy with unidirectional barbed suture — Patients will be randomized to repair of the uterine defect during laparoscopic myomectomy using unidirectional barbed suture material (V-Loc 180TM, CovidienTM). For patients randomized to the barbed suture arm of the trial, any secondary fibroid that is greater than 5cm intra-operatively (as measured by a laparoscopic measurement instrument) will also be closed with barbed suture material. The cut-off of 5cm will be used, since it is generally above this size when uterine defects need to be closed in multiple layers, making the barbed suture potentially useful. Any other secondary fibroids less than 5cm will be closed with traditional extracorporeal suturing in both arms of the trial, since these can usually be closed in one layer.
  Other Names: V-Loc 180TM, CovidienTM
  Arms: Barbed suture
Procedure: Traditional suture material — Patients will be randomized to repair of the uterine defect during laparoscopic myomectomy using traditional extracorporeal suturing using absorbable monofilament suture material.
  Arms: Traditional suture material

SUMMARY:
The objective of this study is to determine if the use of a new type of barbed suture material for laparoscopic myomectomy (surgical removal of fibroids) versus the traditional approach of suturing with conventional suture material to close the uterine defect once the fibroid has been removed, improves surgical outcomes. Specifically, the investigators will investigate the effect of barbed suture on operative time, blood loss, adverse post-operative events and hospital stay.

DETAILED DESCRIPTION:
Although the laparoscopic myomectomy has benefits over the abdominal approach, such as less blood loss, less hemoglobin drop post-operatively, decreased post-operative pain and fewer overall complications, it is a difficult procedure, which often requires greater operative time to perform. In the current climate of attempting to reduce health care expenditures, even though the minimally invasive approach offers the advantage of reduced hospital stay, a deterrent for hospital administration and surgeons may be the increased operative time it may require. Barbed suture is a relatively new material available in gynecologic surgery. Barbs are cut into the suture with the barbs facing in a direction opposite that of the needle. The barbs allow for anchoring of the suture in tissues, which prevents migration and allows suturing without knot tying. This study will be a single-centre non-blinded randomized controlled trial comparing laparoscopic myomectomy with barbed suture versus traditional suture material.

ELIGIBILITY:
Inclusion Criteria:

* women who are planning to undergo laparoscopic myomectomy

Exclusion Criteria:

* greater than five fibroids
* uterus extending beyond the umbilicus
* major medical comorbidity or psychiatric illness, which could affect follow-up and/or compliance
* patients undergoing concomitant surgical procedures at the time of myomectomy (such as resection of endometriosis or ovarian cystectomy)
* pregnancy (all patients will have serum pregnancy testing prior to surgery)
* patients with any suggestion of abnormal pathology on imaging or endometrial biopsy

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2012-01; Primary Completion 2014-01 (Estimated)

PRIMARY OUTCOMES:
Operative time
  We will record the operative time from beginning to completion of suturing each fibroid separately, as well as total operative time for the entire procedure.

SECONDARY OUTCOMES:
Blood loss | Intra-operative
  We will subtract the amount of irrigation fluid used from the total amount of fluid suctioned during the procedure to arrive at an estimated blood loss in millilitres. We will also measure the patient's hemoglobin at the routine pre-operative visit and then on the morning of the first post-operative day to determine the difference in hemoglobin. The amount of intravenous fluids administered to the patients intra- and post-operatively will be documented in order to account for any changes in hemoglobin that are spurious due to fluid administration.
Adverse events | Intra-operatively until 6 weeks post-operatively
  All adverse events that occur until 6 weeks post-operatively will be documented including injury to the bladder, bowel, ureter or blood vessel, infection/abscess, fever, blood transfusion, readmission to hospital, re-operation, and venous thromboembolism.
Hospital stay
  We will document the length of hospital stay post-operatively in days.
Fertility and pregnancy-related outcomes | 2 and 5 years post-operatively
  Telephone interviews will be conducted at 2 and 5 years post-operatively to determine pregnancy rates, live birth rates and adverse pregnancy outcomes of participants.

CONTACTS AND LOCATIONS:
Overall Officials: Jamie Kroft, MD, FRCSC, Principal Investigator — Sunnybrook Health Sciences Centre, University of Toronto; Grace Y Liu, MD, FRCSC, Principal Investigator — Sunnybrook Health Sciences Centre, University of Toronto
Locations (1):
- Sunnybrook Health Sciences Centre, Toronto, Ontario, Canada